CLINICAL TRIAL: NCT07113730
Title: Retrospective and Prospective Study on the Kinetics Profiling of Immune Reconstitution and Clinical Outcomes in CMML Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: The Kinetics Profiling of Immune Reconstitution and Clinical Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Hospital of Jilin University (Other); the 960th Hospital of the People's Liberation Army Joint Logistics Support Force (Unknown); Shanghai General Hospital, ShanghaiJiao Tong University School of Medicine (Unknown)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology Affiliation: Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: 2025PHB073-001
Record Dates: First submitted 2025-07-27; First posted 2025-08-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Myelomonocytic Leukemia (CMML); Immune Reconstitution
Keywords: Chronic Myelomonocytic Leukemia (CMML); immune reconstitution; allogeneic hematopoietic stem cell transplantation (allo-HSCT)
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Immune Reconstitution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective cohort: Patients whose first visit to our institution and the termination of follow-up both occurred before the opening of this study will contribute to the retrospective cohort.
  Interventions: Other: immune reconstitution
- Prospective cohort: Patients whose first visit to our institution occur after the opening of this study will contribute to the prospective cohort.
  Interventions: Other: immune reconstitution
- Retrospective/Prospective cohort: Patients whose first visit to our institution occurred before the opening of this study and whose follow-up will terminate after the opening of this study will contribute to the ambispective cohort.
  Interventions: Other: immune reconstitution

INTERVENTIONS:
Other: immune reconstitution — Detection of immune reconstitution in peripheral blood of patients by flow cytometry at 30-day intervals for 180 days post-transplantation.

SUMMARY:
Chronic myelomonocytic leukemia (CMML) is a clonal hematopoietic malignancy with poor prognosis. Allogeneic hematopoietic stem cell transplantation (HSCT) remains the only potentially curative treatment. Immune reconstitution (IR) is critical for improving HSCT efficacy and quality of life among survivors, yet its dynamic impact on survival and complications like chronic graft-versus-host disease (cGVHD) in CMML is poorly defined. This study aimed to investigate the dynamics of IR following HSCT in patients with CMML and evaluate its impact on post-transplant clinical outcomes.

DETAILED DESCRIPTION:
Chronic myelomonocytic leukemia (CMML) is a myeloid malignancy exhibiting clinical and morphological features of both myelodysplastic syndromes (MDS) and myeloproliferative neoplasms (MPNs). The optimal treatment regimen remains unclear, and allogeneic hematopoietic stem cell transplantation (allo-HSCT) is currently the only known potentially curative treatment option. During allo-HSCT, the recipient's immune system undergoes reconstitution from donor-derived cells. Timely engraftment and functional recovery of the donor immune system are critical for patient recovery and long-term survival post-transplantation. While HSCT can achieve durable remission, it is associated with significant life-threatening complications, primarily mediated by rapidly reconstituted immune components. However, the cellular dynamics underlying the re-establishment of immune homeostasis between donor and recipient compartments post-HSCT remain poorly characterized. This study aims to delineate the kinetics of immune reconstitution (IR) in CMML patients following allo-HSCT, dynamically analyze its impact on clinical outcomes and prognosis, and ultimately develop and optimize immunotherapeutic strategies to enhance overall survival and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of CMML following HSCT
2. Patients treated at Peking University People's Hospital since January 1, 2005

Exclusion Criteria:

1. Any condition that may render follow-up data unreliable, including but not limited to severe psychiatric disorders
2. Patients deemed ineligible for the study by investigators

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed chronic myelomonocytic leukemia (CMML)
  Prerequisite criteria:
  1. persistent of monocytosis in PB (absolute ≥0.5 × 109/L or relative ≥10%)
  2. blast cell <20% in PB and bone marrow, excluding chronic myeloid leukemia or other MPN.
  Supporting criteria :
  1. dysplasia involving 1 or more myeloid lineages
  2. the presence of acquired clonal cytogenetic or molecular abnormalities
  3. abnormal partitioning of PB monocyte subsets (classical monocytes >94%). The requirements for CMML diagnosis include prerequisite criteria that must be met in all patients.
  Then, if the monocyte count is ≥1 × 109/L, one or more supporting criteria must be met, and if the monocyte count is ≥0.5 and <1 × 109/L, the first two supporting criteria must be met.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2035-07-31 (Estimated); Study Completion 2036-07-31 (Estimated)

PRIMARY OUTCOMES:
Immune reconstitution | 180 days
  To quantify the percentages（%） of lymphocyte subsets (including CD19+ B cells, CD3+ T cells, CD4+ T cells, CD8+ T cells, CD3+CD8+CD28+ T cells, CD3+CD4+CD28+ T cells, CD4+CD45RA+ naive T cells, CD4+CD45RO+ memory T cells, CD4+CD25+CD45RA+ naive regulatory T cells, CD4+CD25+CD45RO+ memory regulatory T cells, and CD4+CD25+ total regulatory T cells) relative to nucleated cells using flow cytometry.
Immunoglobulin levels | 180 days
  To test for serum immunoglobulin (IgG, IgA, IgM) (mg/dL).
2-year OS | 2 years
  To describe the incidence of 2-year OS
5-year PFS | 5 years
  To describe the incidence of 5-year PFS

SECONDARY OUTCOMES:
cGVHD | 5 years
  To describe the number of patients diagnosed with chronic graft-versus-host disease (cGVHD)
Bacterial infection | 5 years
  To describe the number of patients with bacterial infection detected in blood, stool, sputum, etc. after HSCT
Fungal infection | 5 years
  To describe the number of patients with fungal infection detected in blood, stool, sputum, etc. after HSCT
Viral infection | 5 years
  To describe the number of patients with viral infection detected in blood, stool, sputum, etc. after HSCT
aGVHD | 100 days
  To describe the number of patients diagnosed with acute graft-versus-host disease (aGVHD)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital